CLINICAL TRIAL: NCT02978976
Title: The Effect of Maternal Antenatal Steroid Administration on the Blood Flow Through the Pulmonary Artery in the Term Fetus; a Randomized Control Double Blinded Study
Brief Title: Effect of Antenatal Steroid on Pulmonary Artery Blood Flow
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer of Obstetrtics & gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A22102016
Record Dates: First submitted 2016-10-22; First posted 2016-12-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Neonatal Respiratory Distress
Keywords: RDS; Doppler on fetal pulmonary artery
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Betamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- betamethasone (Experimental): will receive two doses of 12mg betamethasone, then the pulsatility index (PI), resistance index (RI), systolic/diastolic ratio (SD), and the acceleration-time/ejection-time ratio (At/Et) will be determined in all cases after recruitment, just before the administration of the drug (betamethasone), 24 hours after the last dose, and on the day of elective Cs.
  Interventions: Drug: Betamethasone
- Saline (Placebo Comparator): will receive saline injection placebo, then the pulsatility index (PI), resistance index (RI), systolic/diastolic ratio (SD), and the acceleration-time/ejection-time ratio (At/Et) will be determined in all cases after recruitment, just before the administration of the drug ( placebo), 24 hours after the last dose, and on the day of elective Cs.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Betamethasone — will receive two doses of 12mg betamethasone ( Dipropfos ® SCHERING-PLOUGH; Kenilworth, New Jersey, USA) intramuscularly (IM) 24 hours apart.
  Other Names: Dipropfos
  Arms: betamethasone
Drug: saline — saline placebo injection in the same regimen.
  Other Names: NaCl 0.9
  Arms: Saline

SUMMARY:
The aim of this study is to determine the effect of administering antenatal steroids in term fetuses on the blood flow in the fetal pulmonary artery, and to correlate these findings with clinical data obtained after birth documenting respiratory disorders.

DETAILED DESCRIPTION:
After internal review board approval, 126 consecutive patients attending the antenatal care clinic of Kasr Alainy Hospital, part of Cairo university hospitals will be recruited in this study. All patients will sign informed consent.

Patients included in the study will be 20-38 years of age, have an indication for elective caesarean section. Patients will be excluded if they are hypertensive, diabetic or have any disorder that may be aggravated by administration of steroids, women with systemic infection including tuberculosis or sepsis, any fetal congenital anomalies (affecting the fetal heart, lungs, and circulation), history of rupture membranes, or suspected chorioamnionitis, intrauterine growth retardation (IUGR), and intrauterine fetal demise (IUFD).

Patients will be randomized on 37 weeks and 6 days gestation by the nurse attending the clinic using a computer generated randomization table, and a closed envelope system will be used. Patients will be equally divided into two groups. Patients in group (A) will receive two doses of 12mg betamethasone ( Dipropfos ® SCHERING-PLOUGH; Kenilworth, New Jersey, USA) intramuscularly (IM) 24 hours apart, while group (B) patients will receive a saline placebo injection in the same regimen.

Ultrasound examination will be done where all patients will lie down in a semi-recumbent position, and the ultrasound will be performed by an expert ultrasonographer, with expert training in fetal echocardiography. The ultrasound specialist will be blinded to which study arm the patients belongs. The abdominal probe of the ultrasound machine (voluson730; kretz,Zipf,Austria) will be placed so that the fetal chest will be in a transverse section, giving us the four chamber view of the fetal heart. The color Doppler will then be switched on, and the fetal pulmonary artery will be identified. The measurements will be taken from the middle segment of the pulmonary artery just after the first bifurcation of the pulmonary branch (just after crossing the aortic arch). We will obtain our measurements from either the right or left pulmonary arteries, whichever is easier according to fetal position, as there is no difference between the values obtained from either according to the work done by Rasanen et al.

The pulsatility index (PI), resistance index (RI), systolic/diastolic ratio (SD), and the acceleration-time/ejection-time ratio (At/Et) will be determined in all cases after recruitment, just before the administration of the drug (betamethasone / placebo), 24 hours after the last dose, and on the day of elective Cs. Caesarean section will be performed 7 days after the last dose of betamethasone, and a senior neonatologist will attend the birth, document Apgar score, and any neonatal respiratory distress.

A sample size was calculated where the difference in the mean pulsatility index (PI) before and after administration of antenatal steroids for the middle segment of the fetal pulmonary artery was 0.42 in a previous study by Bartha et al, and the standard deviation was set as 0.79. The Type I error probability was set at 0.05, and the power at 80%. This gave us 57 patients in each arm, and allowing for dropout rate of 10%, 63 patients will be recruited in each arm of the study, as the ratio between both study and control was 1:1. PS Power and Sample size Calculations software, Versionv2.1.30 for MS Windows, was used to calculate sample size Dupont and Vanderbilt, USA).

ELIGIBILITY:
Inclusion Criteria:

* indication for elective caesarean section.
* 37weeks +6days

Exclusion Criteria:

* hypertensive
* diabetic
* any disorder that may be aggravated by administration of steroids
* women with systemic infection including tuberculosis or sepsis
* any fetal congenital anomalies (affecting the fetal heart, lungs, and circulation)
* history of rupture membranes, or suspected chorioamnionitis
* intrauterine growth retardation (IUGR)
* intrauterine fetal demise (IUFD).

Ages: 28 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
changes in the mean doppler parameters between the study groups before and after the drug administration ( compare means of doppler reading between both groups using t-test) | 1 week

SECONDARY OUTCOMES:
Presense of respiratory disorders in neonate (yes/no) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamel, M.D., Principal Investigator — Lecturer Of obstetrics and gynecology
Locations (1):
- 11562, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
yes

REFERENCES:
- [Background] Bartha JL, Largo-Heinrich M, Machado MJ, Gonzalez-Bugatto F, Hervias-Vivancos B. Effects of antenatal betamethasone on human fetal branch pulmonary artery flow velocity waveforms. Fetal Diagn Ther. 2008;23(1):46-53. doi: 10.1159/000109226. Epub 2007 Oct 9. PMID 17934298